CLINICAL TRIAL: NCT03000335
Title: Evaluation of ProALL microRNAs in Blood Specimen for Prediction of Acute Lymphoblastic Leukemia Relapse Risk
Brief Title: Evaluation of ProALL miRs in Blood Specimen for Prediction of ALL Relapse Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Curewize Health Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CW003
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: microRNA; relapse; blood; in vitro diagnostics; prediction; lab test
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples will be collected and transcribed to RNA. RNA samples will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Relapse: B-ALL patients who have succumbed to relapse
- Remission: B-ALL patients who are in remission

SUMMARY:
Previous findings have shown that a biomarker comprised of the three microRNAs (miRs) miR-451, miR-151-5p and miR-1290 can independently predict precursor B-cell acute lymphoblastic leukemia (B- ALL) patients' risk for relapse when measured in cells from a bone marrow (BM) aspiration taken at diagnosis (Avigad et al., 2016: Genes, Chromosomes & Cancer 55:328-339). Curewize Health recognizes that the development of a minimally invasive blood test for frequent long-term monitoring can greatly benefit pediatric precursor B-ALL patients. Therefore, the current study will investigate the monitoring ability of miR-451, miR-151-5p and miR-1290 measured in blood samples. The study will be performed in two stages:

Stage 1-Cross-Sectional Study: Blood samples will be collected from relapsed pediatric B-ALL patients and B-ALL patients in remission. Blood will be collected from each patient in three tubes, for serum, plasma and whole blood analysis, in order to interpret the best blood source for measuring miR-451, miR-151-5p and miR-1290. The level of the miRs in blood will be compared between relapsed B-ALL patients to B-ALL patients in remission. If the Stage 1 Cross-Sectional study is successful, the investigators will continue the clinical trials to the Stage 2 Prospective Monitoring study.

Stage 2-Prospective Monitoring Study: Blood will be collected from patients at diagnosis and at routine clinical follow-up. Patients can be up to five years from diagnosis. The source of blood found to be most optimal for measuring the miR levels is Stage 1 will be collected. The final design of the Stage 2 study will be decided after completion of the Stage 1 study.

DETAILED DESCRIPTION:
1. Acute Lymphoblastic Leukemia Risk Based Treatment:

   Children with ALL are usually treated according to risk groups defined by both clinical and laboratory features. This approach allows children with signs of historically very good outcome to be treated with modest therapy and to be spared more intensive and toxic treatment, while allowing children with a historically lower probability of long-term survival to receive more intensive therapy that may increase the ALL patients' chance of cure. Study groups use varying criteria, with a strong emphasis on minimal residual disease (MRD) measurements that quantify the number of leukemic cells that remain in the patient during and after treatment. The most widely used MRD assays are based on polymerase chain reaction (PCR) amplification of antigen-receptor genes, and on flow cytometric detection of abnormal immunophenotypes (Campana, 2010). These techniques identify the patients' specific leukemia clone in bone marrow before induction treatment and measure the number of residual leukemic cells post-induction. Two widely used examples of Risk stratification protocols are the Berlin-Frankfurt-Munster (BFM) Protocol in Europe and the Children's Oncology Group Protocol in USA.
2. Previous ProALL miR Findings:

   The ProALL prototype assay microRNAs (miRNAs) (Avigad et al., 2016) were discovered by microarray analysis by hybridization of BM aspirates taken at diagnosis of 48 ALL patients to 979 different miRNAs. The down-regulated expression levels of miR-451 and miR-151-5p and the up-regulated expression level of miR-1290 associated with adverse prognostic factors.

   The second study focused on measuring the three miRs in BM samples taken from B-ALL patients at diagnosis treated by the BFM protocol. ProALL miRs predicted high risk to relapse (p<0.0001, n=127). ProALL miRs were found to be an independent predictor when tested with prognostic factors known at diagnosis and when tested with PCR-MRD. Similar findings were found for patients treated by the DCOG protocol (n=32, p<0.0001). In a small feasibility study the investigators showed that ProALL miRs measured in blood correlated with ProALL miRs measured in bone marrow (Avigad et al. Mir Expression Profile of Peripheral Blood Lymphocytes Predicts Relapse in Pediatric Acute Lymphoblastic Leukemia. Blood. 2016;128:1736 - Poster presentation at ASH 2016).
3. Study Rationale:

   Though MRD has greatly contributed to the substantial increase in ALL patients' survival and outcome, nearly 15% to 20% of young ALL patients eventually succumb to relapse, resulting in relapsed ALL as being the 4th most common childhood malignancy (Locatelli et al., 2012, Pui et al., 2012, Hunger and Mullighaan, 2015). Once relapse occurs only 30% to 50% of relapsed patients can be cured even with intensive chemotherapy and bone marrow transplantation (Nguyen et al. 2008 and Locatelli et al., 2012). Relapsed ALL patients with high MRD prior to hematopoietic stem cell transplantation (HSCT) have a significantly worse probability of disease-free survival 10 years after relapse treatment begins (Eckert et al., 2015). Therefore, it stands to reason that early detection of relapse before a large increase in MRD can improve relapse patients disease-free survival. Yet, many oncology groups don't incorporate monitoring in ALL treatment protocols because of the labor intensity of MRD measurement; and the invalidation of the feasibility of routine MRD monitoring. This is due to factors such as variable kinetics of leukemic cell regrowth (van Dongen et al., 2015), and that nearly 50% of ALL patients succumb to relapse from a new leukemia clone not identified at diagnosis (Choi et al., 2007). The frequency of monitoring may also be limited, especially in children, due to discomfort and practical difficulties posed by BM aspiration (Coustan-Smith E. et al., 2002). A simple predictive test for ALL in blood would increase the practicality of testing ALL patients more frequently and may eventually lead to prevention of relapse by means of preemptive treatment.

   Investigating if ProALL miRs can be measured in blood, in addition to BM, for predicting relapse risk of ALL patients is vital due to the many advantages of such a blood test. If ProALL levels can be tested more frequently in blood the probability of successfully treating the patients' leukemia will increase by potentially enabling the physician to take preemptive measures to prevent predicted relapse.
4. Study Design:

   The study will be performed in two stages:

   Stage 1-Cross-Sectional Study: Blood samples will be collected from relapsed pediatric B-ALL patients and B-ALL patients in remission. Three Blood samples will be collected from each patient in tubes in order to interpret the best blood source for measuring miR-451, miR-151-5p and miR-1290. The sources that will be tested are serum, peripheral blood lymphocytes and whole blood. The level of the miRs in blood will be compared between relapsed B-ALL patients and B-ALL patients in remission (n=30). If the "Stage 1 Cross-Sectional" study is successful, the investigators will continue the clinical trial to the "Stage 2 Prospective Monitoring" study.

   Stage 2-Prospective Monitoring Study: Blood will be collected from patients at diagnosis and/or at routine clinical follow-up. Patients can be up to five years from diagnosis (n≈65 *3 samples). One source of blood will be collected. Patients will be followed for 3 years. The final design of the Stage 2 study will be after the completion of Stage 1 study.
5. Sample Size Considerations:

   Stage 1 Cross-Sectional Study: For the sample size calculation the Primary end-point is to test the ability of ProALL miRs measured in blood to differentiate B-ALL patients at remission from patients at relapse. The sample size calculation is according to Sampling: comparison of proportions of MedCalc (MedCalc Statistical Software version 16.1 (MedCalc Software bvba, Ostend, Belgium; https://www.medcalc.org; 2016). Type 1 error was 0.05 and Type 2 error was 0.20. Data for the sample size calculation was obtained from the DCOG cohort in Avigad et al., 2016, which was chosen as a model for the feasibility study due to its small size (n=32). Cross sectional analysis of the DCOG cohort showed that there were significantly more patients with relapse event (p=0.001, Fisher Exact test) positive for at least one miR (78%) compared to patients with no relapse event (13%).

   Data is taken from Figure 6 (from Avigad et al., 2016):
   * Patients at Relapse - At least one miR positive rate 0.78
   * Patients at Remission - No miR positive rate 0.13
   * Relapse/Remission was 0.39
   * The minimum number of enrollees needed are: a. Patients at Relapse - n=8 and b. Patients at Remission - n=21.

   B-ALL patients can be included in the study up to five years from diagnosis. After completing the enrollment of the cross-sectional study, PI will be queried on Remission/Relapse status of patients. Above is the minimum number of patients to be enrolled. Up to 12 patients at relapse and 31 patents at remission can be enrolled.

   Stage 2 Prospective Study: The sample size calculation is according to Sampling: survival analysis (Time-to-Event) of MedCalc. Type 1 error was 0.05 and Type 2 error was 0.20. Data for the sample size calculation was obtained from Figure 3A Kaplan Meir curve (Avigad et al., 2016).
   * Survival rate Profile B was 0.77
   * Survival rate Profile A was 0.29
   * Profile B/Profile A was 17
   * Number of enrollees needed is 62

   At least 3 samples from 3 time points should be taken from each patient. A sample can be taken at relapse if it is the 2nd or 3rd sample. Patients from Stage 1 can continue to Stage 2. The final design of the study will be after Stage 1.
6. Blood Extraction and Handling of Samples:

   No more than 0.8 mL of blood per kilogram of the enrollee's weight will be collected at one visit. The total amount of blood to be collected for Stage 1 is between 7.5 mL to 10.5 mL according to the following:.
   * PaxGene Tube - 2.5 mL
   * Tube for Plasma - 2.5 mL to 4 mL
   * Tube for Serum - 2.5 mL to 4 mL
7. Biomarker Results and Clinical Data Flow:

   * The blood samples will be screened for the ProALL miRs by Curewize Lab.
   * Curewize will receive clinical data corresponding to the visit that the screened blood sample was taken only after sending the clinical site the blood sample's miR values.
8. Statistical Analysis Plan (SAP) for Stage 1-Cross Sectional Study:

   Blood Biomarker Variables:
   * miR-451 relative expression (ddCt) level
   * miR-151-5p relative expression (ddCt) level
   * miR-1290 relative expression (ddCt) level

   Covariates:
   * Age
   * Gender
   * MRD-PCR
   * BFM risk
   * Treatment group
   * White blood cell count at diagnosis and at blood collection if routinely tested.
   * Steroid response
   * Cytogenetic variables

   Cross-Sectional Analysis:

   Stage-1 is considered exploratory and will be used to design the analysis of Stage-2.

   Variables will be tested for normality with Shapiro Wilk's test. The level of expression of miR-451, miR151-5p and miR-1290 will be compared between patients during remission and patients during relapse by Mann-Whitney U test. Continuous data will be depicted in box plots showing median and interquartile range. Logistic regression will be used to test the miR values [nominal (positive/negative) and continuous] with each other and with other variables comparing between patients at remission and patients at relapse. The optimal combination Classifier will be created according to the above analysis. Categorical variables will be summarized by frequency tables, indicating numbers and frequencies of miR status (positive versus negative). Data will be compared by Fisher exact for dichotomous (2x2 tables) values or chi-square or chi-square for trend for tables. Odds ratios and likelihood ratios will be calculated. Receiver operating characteristic curves will be created, the independent variables are miR-451 or miR-151-p, miR-1290 and dependent variable is relapse or remission. Receiver operating characteristic curves will be created for the combined Classifier. Additional analyses will be performed if results from planned analyses give reasonable warrant.
9. Statistical Analysis Plan (SAP) for Stage 2-Prospective Study Will be created after report of results of Stage-1 Cross Section Study.
10. Ethical Considerations The study will be conducted according to the principles of the World Medical Association Declaration of Helsinki Ethical Principles for Medical Research Involving Human Subjects JAMA. 2013;310(20):2191-2194 and in accordance with local GCP regulations.

ELIGIBILITY:
Inclusion Criteria:

* Written inform consent was given for the clinical trial by the subject or subject's legally acceptable representative.
* Patient with a final diagnosis of B-ALL
* Male or Female
* Age from 2 to 19 years at diagnosis.
* Patient during remission at least 3 months after starting treatment.
* Patient is up to five years from diagnosis at the baseline visit.
* Patient at relapse before starting treatment for relapse.
* Patient weighs at least 9.4 kg.

Exclusion Criteria:

* Discovery of an alternative disorder other than B-cell acute lymphoblastic leukemia.
* The subject has known human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibody or other dangerous contagious disease.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * B-ALL patients at relapse
  * B-ALL patients at remission
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Abilty of miR-451, miR-151-5p and miR-1290 to Differentiate B-ALL Patients in Relapse from Patients in Remission | Maximum One and half years after enrollment of first patient
  Investigate the ability of miR-451, miR-151-5p and miR-1290 measured in blood samples to differentiate between B-ALL patients who are in remission to patients who are in relapse.
Stage 2: Ability of miR-451, miR-151-5p and miR-1290 to Monitor B-ALL Patients | Three and a half years from enrollment of first patient
  Investigate the ability of miR-451, miR-151-5p and miR-1290 measured in blood samples as a surveillance monitoring tool to detect molecular relapse before overt clinical relapse and to confirm sustained molecular remission.

SECONDARY OUTCOMES:
Stage 1: Optimal Blood Source for Measuring miR-451, miR-151-5p and miR-1290 for Monitoring B-ALL Patients | Maximum One and half years after enrollment of first patient
  Investigate the optimal source of blood for the measurement of miR 451, miR-151-5p and miR-1290 for monitoring B-ALL patients for molecular relapse before overt clinical relapse and confirm sustained molecular remission.
Stage 1: Decide if to Continue to Stage 2 Prospective Monitoring Study of the three miRs. | Maximum One and half years after enrollment of first patient
  If results from Outcome 1 are positive then the study will continue to Stage 2.
Stage 1: Finalize the design of Stage 2 Prospective Monitoring Study. | Maximum One and half years after enrollment of first patient
  Sample size considerations and design of Stage 2 of the study will be finalized according to results of Stage 1.
Stage 2: Combined Classifier for Monitoring B-ALL Patients for Overt Clinical Relapse or Sustained Remission | Four years from enrollment of first patient
  Develop ProALL monitoring classifier based on the measurement of miR-451, miR 151-5p and miR-1290 in blood. An algorithm will be created that includes the most optimal combination and level changes of the microRNA to use as a surveillance monitoring tool of B-ALL patients.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Yaniv, MD, Study Chair — Schneider Children's Medical Center, Israel
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckert C, Hagedorn N, Sramkova L, Mann G, Panzer-Grumayer R, Peters C, Bourquin JP, Klingebiel T, Borkhardt A, Cario G, Alten J, Escherich G, Astrahantseff K, Seeger K, Henze G, von Stackelberg A. Monitoring minimal residual disease in children with high-risk relapses of acute lymphoblastic leukemia: prognostic relevance of early and late assessment. Leukemia. 2015 Aug;29(8):1648-55. doi: 10.1038/leu.2015.59. Epub 2015 Mar 9. PMID 25748682
- [Background] Choi S, Henderson MJ, Kwan E, Beesley AH, Sutton R, Bahar AY, Giles J, Venn NC, Pozza LD, Baker DL, Marshall GM, Kees UR, Haber M, Norris MD. Relapse in children with acute lymphoblastic leukemia involving selection of a preexisting drug-resistant subclone. Blood. 2007 Jul 15;110(2):632-9. doi: 10.1182/blood-2007-01-067785. Epub 2007 Mar 19. PMID 17371950
- [Background] Coustan-Smith E, Sancho J, Hancock ML, Razzouk BI, Ribeiro RC, Rivera GK, Rubnitz JE, Sandlund JT, Pui CH, Campana D. Use of peripheral blood instead of bone marrow to monitor residual disease in children with acute lymphoblastic leukemia. Blood. 2002 Oct 1;100(7):2399-402. doi: 10.1182/blood-2002-04-1130. PMID 12239148
- [Background] Hunger SP, Mullighan CG. Redefining ALL classification: toward detecting high-risk ALL and implementing precision medicine. Blood. 2015 Jun 25;125(26):3977-87. doi: 10.1182/blood-2015-02-580043. Epub 2015 May 21. PMID 25999453
- [Background] Locatelli F, Schrappe M, Bernardo ME, Rutella S. How I treat relapsed childhood acute lymphoblastic leukemia. Blood. 2012 Oct 4;120(14):2807-16. doi: 10.1182/blood-2012-02-265884. Epub 2012 Aug 15. PMID 22896001
- [Background] Nguyen K, Devidas M, Cheng SC, La M, Raetz EA, Carroll WL, Winick NJ, Hunger SP, Gaynon PS, Loh ML; Children's Oncology Group. Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia. 2008 Dec;22(12):2142-50. doi: 10.1038/leu.2008.251. Epub 2008 Sep 25. PMID 18818707
- [Background] Pui CH, Mullighan CG, Evans WE, Relling MV. Pediatric acute lymphoblastic leukemia: where are we going and how do we get there? Blood. 2012 Aug 9;120(6):1165-74. doi: 10.1182/blood-2012-05-378943. Epub 2012 Jun 22. PMID 22730540
- [Result] Avigad S, Verly IR, Lebel A, Kordi O, Shichrur K, Ohali A, Hameiri-Grossman M, Kaspers GJ, Cloos J, Fronkova E, Trka J, Luria D, Kodman Y, Mirsky H, Gaash D, Jeison M, Avrahami G, Elitzur S, Gilad G, Stark B, Yaniv I. miR expression profiling at diagnosis predicts relapse in pediatric precursor B-cell acute lymphoblastic leukemia. Genes Chromosomes Cancer. 2016 Apr;55(4):328-39. doi: 10.1002/gcc.22334. Epub 2015 Dec 19. PMID 26684414
- See also: Sponsor — http://www.curewize.com